CLINICAL TRIAL: NCT03078816
Title: Thalamic Deep Brain Stimulation for Secondary Dystonia in Children and Young Adults
Acronym: DBSVop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 123822A
Record Dates: First submitted 2016-04-26; First posted 2017-03-13 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- DBS active (Experimental): All participants will be enrolled in DBS placement and active stimulation. The following components will be used:
  * Activa PC Primary Cell Neurostimulator - (Model 37601)
  * Activa RC Rechargeable Neurostimulator - (Model 37612)
  * Activa SC Single Cell Neurostimulator (Models 37602 and 37603)
  * DBS Lead - (Model 3387)
  * DBS Extension - (Models 37085/6)
  * Patient Programmer - (Model 37642)
  * Test Stimulator - (Model 3625)
  * N'Vision Clinician Programmer - (Model 8840)
  * N'Vision Software Application Card - (Model 8870)
  Interventions: Device: Activa PC Primary Cell Neurostimulator - (Model 37601); Device: Activa RC Rechargeable Neurostimulator - (Model 37612); Device: Activa SC Single Cell Neurostimulator (Models 37602/37603); Device: DBS Lead - (Model 3387; Device: DBS Extension - (Models 37085/6); Device: Patient Programmer - (Model 37642); Device: Test Stimulator - (Model 3625); Device: N'Vision Clinician Programmer - (Model 8840); Device: N'Vision Software Application Card - (Model 8870)

INTERVENTIONS:
Device: Activa PC Primary Cell Neurostimulator - (Model 37601) — Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.
Device: Activa RC Rechargeable Neurostimulator - (Model 37612) — Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.
Device: Activa SC Single Cell Neurostimulator (Models 37602/37603) — Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.
Device: DBS Lead - (Model 3387 — Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.
Device: DBS Extension - (Models 37085/6) — Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.
Device: Patient Programmer - (Model 37642) — Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.
Device: Test Stimulator - (Model 3625) — Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.
Device: N'Vision Clinician Programmer - (Model 8840) — Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.
Device: N'Vision Software Application Card - (Model 8870) — Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.

SUMMARY:
Dystonia is a movement disorder seen in both children and adults that is characterized by "sustained or intermittent muscle contractions causing abnormal, often repetitive, movements, postures, or both." Secondary dystonia is far more common in pediatric populations than primary dystonia, and far more recalcitrant to standard pharmacologic and surgical treatments including Deep Brain Stimulation (DBS). There exists a large unmet need to develop new therapeutics, treatment strategies, and outcome measures for pediatric secondary dystonia.

The investigators are proposing to investigate the ventralis oralis posterior nucleus (Vop) of the thalamus as a new target for DBS in secondary dystonia. Prior to the development of DBS, the main surgical treatment of dystonia was thalamotomy. Although there were many different targets in the thalamus, often done in staged procedures, the most common and successful targeted nuclei was the Vop, which is traditionally thought to be the pallidal receiving area. Previous lesioning of Vop produced improvements in dystonia but intolerable side effects, especially when implanted bilaterally. However, given that secondary dystonia patients were often reported to have superior results to primary dystonia it is reasonable to believe that if the side effects can be modulated, that targeting of the Vop nucleus with DBS could be a viable alternative to Globus Pallidus interna (GPi). Given that Deep Brain Stimulation is a treatment that is inherently adjustable, it is conceivable that settings on the Deep Brain Stimulation could be adjusted to allow for clinical benefit with minimal side effects. Indeed, there have been several scattered successful case reports attesting to this possibility.

DETAILED DESCRIPTION:
Dystonia is a movement disorder seen in both children and adults that is characterized by "sustained or intermittent muscle contractions causing abnormal, often repetitive, movements, postures, or both." Secondary dystonia has evolved to refer to dystonia resulting from damage to the nervous system or degenerative disease processes. While primary dystonia is generally thought to arise from genetic causes, secondary dystonias have a variety of causes including perinatal injuries (cerebral palsy), central nervous system infections, traumatic brain injuries, and many different metabolic, neurodegenerative, and mitochondrial conditions. Secondary dystonia is far more common in pediatric populations than primary dystonia, and far more recalcitrant to standard pharmacologic and surgical treatments including Deep Brain Stimulation. Given that most treatments for dystonia are developed for primary dystonia and then applied to secondary dystonia, it is not surprising that this effectiveness gap exists. Thus, there exists a large unmet need to develop new therapeutics, treatment strategies, and outcome measures for pediatric secondary dystonia.

Deep Brain Stimulation (DBS) is one such therapeutic intervention that has potential to improve secondary dystonia. DBS is a surgical treatment for several different movement disorders that evolved from functional stereotactic neurosurgery techniques initially used to lesion specific deep brain structures. While Essential Tremor and Idiopathic Parkinson's Disease have predictable and consistent response rates to DBS in carefully selected patients, response rates of dystonia have been much more inconsistent. One predictor of success has been the presence of DYT-1 mutation, the most common known genetic cause of primary dystonia. Success rates in DYT-1 dystonia are consistently high with reductions in dystonia typically greater than 80%. However, the results in secondary dystonia have been much more modest and inconsistent. A recent meta-analysis found that on average, dystonia symptoms as measured by common rating scales improve 23% following DBS for dystonic cerebral palsy (the most common cause of secondary dystonia), however there are frequent cases of non-responders. Additionally, there have been very few examination, radiological or laboratory predictors of good response to DBS, except for genetic confirmation of DYT-119. However, across both primary and secondary dystonia, younger age at the time of surgery (less than 21 years old) and shorter duration of symptoms (less than 15 years) have been shown to be the most likely predictive factors for a good postoperative outcome. This has led many to suggest that DBS should be offered earlier in the course of intractable dystonia, prior to the development of permanent complications such as orthopedic contractures. Thus, we are setting an upper age limit of 25 to account for the concern that earlier implantation leads to improved outcomes. The lower age limit of 7 reflects the fact that the current humanitarian exemption for DBS for dystonia currently goes down to age 7. Thus, there exists a need to both improve patient selection as well as application of DBS for secondary dystonia in children.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent or assent for the study
2. Dystonia symptoms that are sufficiently severe, in spite of best medical therapy, to warrant surgical implantation of deep brain stimulators according to standard clinical criteria
3. Age 7-25
4. Stable doses of anti-dystonia medications (such as levodopa, baclofen, or diazepam) for at least 30 days prior to baseline assessment
5. If patient receives botulinum toxin injections, patient should be on a stable injection regimen
6. Intact thalamic anatomy as determined by standard clinical MRI

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Major comorbidity increasing the risk of surgery (severe hypertension, severe diabetes, or need for chronic anticoagulation other than aspirin)
3. Inability to comply with study follow-up visits
4. Any prior intracranial surgery
5. Uncontrolled epilepsy
6. Immunocompromised
7. Has an active infection
8. Requires diathermy, electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) to treat a chronic condition
9. Has an existing implanted neurostimulator or cardiac pacemaker.
10. Dystonia caused by known genetic mutation in any DYT genes

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta San Luciano Palenzuela, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mink JW. Special concerns in defining, studying, and treating dystonia in children. Mov Disord. 2013 Jun 15;28(7):921-5. doi: 10.1002/mds.25548. PMID 23893449
- [Background] Sironi VA. Origin and evolution of deep brain stimulation. Front Integr Neurosci. 2011 Aug 18;5:42. doi: 10.3389/fnint.2011.00042. eCollection 2011. PMID 21887135
- [Background] Franzini A, Cordella R, Messina G, Marras CE, Romito LM, Albanese A, Rizzi M, Nardocci N, Zorzi G, Zekaj E, Villani F, Leone M, Gambini O, Broggi G. Targeting the brain: considerations in 332 consecutive patients treated by deep brain stimulation (DBS) for severe neurological diseases. Neurol Sci. 2012 Dec;33(6):1285-303. doi: 10.1007/s10072-012-0937-9. Epub 2012 Jan 24. PMID 22271259
- [Background] Panov F, Gologorsky Y, Connors G, Tagliati M, Miravite J, Alterman RL. Deep brain stimulation in DYT1 dystonia: a 10-year experience. Neurosurgery. 2013 Jul;73(1):86-93; discussion 93. doi: 10.1227/01.neu.0000429841.84083.c8. PMID 23615098
- [Background] Cif L, Vasques X, Gonzalez V, Ravel P, Biolsi B, Collod-Beroud G, Tuffery-Giraud S, Elfertit H, Claustres M, Coubes P. Long-term follow-up of DYT1 dystonia patients treated by deep brain stimulation: an open-label study. Mov Disord. 2010 Feb 15;25(3):289-99. doi: 10.1002/mds.22802. PMID 20063427
- [Background] Air EL, Ostrem JL, Sanger TD, Starr PA. Deep brain stimulation in children: experience and technical pearls. J Neurosurg Pediatr. 2011 Dec;8(6):566-74. doi: 10.3171/2011.8.PEDS11153. PMID 22132914
- [Background] Koy A, Hellmich M, Pauls KA, Marks W, Lin JP, Fricke O, Timmermann L. Effects of deep brain stimulation in dyskinetic cerebral palsy: a meta-analysis. Mov Disord. 2013 May;28(5):647-54. doi: 10.1002/mds.25339. Epub 2013 Feb 13. PMID 23408442
- [Background] Vidailhet M, Jutras MF, Grabli D, Roze E. Deep brain stimulation for dystonia. J Neurol Neurosurg Psychiatry. 2013 Sep;84(9):1029-42. doi: 10.1136/jnnp-2011-301714. Epub 2012 Nov 15. PMID 23154125
- [Background] Hyam JA, Owen SL, Kringelbach ML, Jenkinson N, Stein JF, Green AL, Aziz TZ. Contrasting connectivity of the ventralis intermedius and ventralis oralis posterior nuclei of the motor thalamus demonstrated by probabilistic tractography. Neurosurgery. 2012 Jan;70(1):162-9; discussion 169. doi: 10.1227/NEU.0b013e3182262c9a. PMID 22158304
- [Background] Andrew J, Fowler CJ, Harrison MJ. Stereotaxic thalamotomy in 55 cases of dystonia. Brain. 1983 Dec;106 ( Pt 4):981-1000. doi: 10.1093/brain/106.4.981. PMID 6360306
- [Background] Burchiel KJ. Thalamotomy for movement disorders. Neurosurg Clin N Am. 1995 Jan;6(1):55-71. PMID 7696875
- [Background] Cardoso F, Jankovic J, Grossman RG, Hamilton WJ. Outcome after stereotactic thalamotomy for dystonia and hemiballismus. Neurosurgery. 1995 Mar;36(3):501-7; discussion 507-8. doi: 10.1227/00006123-199503000-00009. PMID 7753350
- [Background] Kim JP, Chang WS, Chang JW. The long-term surgical outcomes of secondary hemidystonia associated with post-traumatic brain injury. Acta Neurochir (Wien). 2012 May;154(5):823-30. doi: 10.1007/s00701-012-1306-4. Epub 2012 Feb 27. PMID 22367408
- [Background] Vidailhet M, Yelnik J, Lagrange C, Fraix V, Grabli D, Thobois S, Burbaud P, Welter ML, Xie-Brustolin J, Braga MC, Ardouin C, Czernecki V, Klinger H, Chabardes S, Seigneuret E, Mertens P, Cuny E, Navarro S, Cornu P, Benabid AL, Le Bas JF, Dormont D, Hermier M, Dujardin K, Blond S, Krystkowiak P, Destee A, Bardinet E, Agid Y, Krack P, Broussolle E, Pollak P; French SPIDY-2 Study Group. Bilateral pallidal deep brain stimulation for the treatment of patients with dystonia-choreoathetosis cerebral palsy: a prospective pilot study. Lancet Neurol. 2009 Aug;8(8):709-17. doi: 10.1016/S1474-4422(09)70151-6. Epub 2009 Jul 1. PMID 19576854
- [Background] Binder DK, Rau GM, Starr PA. Risk factors for hemorrhage during microelectrode-guided deep brain stimulator implantation for movement disorders. Neurosurgery. 2005 Apr;56(4):722-32; discussion 722-32. doi: 10.1227/01.neu.0000156473.57196.7e. PMID 15792511
- [Background] Sillay KA, Larson PS, Starr PA. Deep brain stimulator hardware-related infections: incidence and management in a large series. Neurosurgery. 2008 Feb;62(2):360-6; discussion 366-7. doi: 10.1227/01.neu.0000316002.03765.33. PMID 18382313
- [Background] Horisawa S, Ochiai T, Goto S, Nakajima T, Takeda N, Fukui A, Hanada T, Kawamata T, Taira T. Safety and long-term efficacy of ventro-oral thalamotomy for focal hand dystonia: A retrospective study of 171 patients. Neurology. 2019 Jan 22;92(4):e371-e377. doi: 10.1212/WNL.0000000000006818. Epub 2018 Dec 26. PMID 30587520
- [Derived] San Luciano M, Robichaux-Viehoever A, Dodenhoff KA, Gittings ML, Viser AC, Racine CA, Bledsoe IO, Watson Pereira C, Wang SS, Starr PA, Ostrem JL. Thalamic deep brain stimulation for acquired dystonia in children and young adults: a phase 1 clinical trial. J Neurosurg Pediatr. 2020 Nov 27;27(2):203-212. doi: 10.3171/2020.7.PEDS20348. Print 2021 Feb 1. PMID 33254134

RESULTS

PARTICIPANT FLOW:
Groups:
- DBS Active: Participants will have DBS placement and active stimulation.The following components will be used:
  * Activa PC Primary Cell Neurostimulator(Model 37601)
  * Activa RC Rechargeable Neurostimulator(Model 37612)
  * Activa SC Single Cell Neurostimulator(Models 37602 and 37603)
  * DBS Lead(Model 3387)
  * DBS Extension(Models 37085/6)
  * Patient Programmer(Model 37642)
  * Test Stimulator(Model 3625)
  * N'Vision Clinician Programmer(Model 8840)
  * N'Vision Software Application Card(Model 8870) Activa PC Primary Cell Neurostimulator(Model 37601): Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.
  Activa RC Rechargeable Neurostimulator - (Model 37612): Deep Brain Stimulator system will be implanted using standard neurosurgical techniques.
Period: Overall Study
Arm/Group | DBS Active
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- DBS Active: All participants will be enrolled in DBS placement and active stimulation. The following components will be used:
  * Activa PC Primary Cell Neurostimulator - (Model 37601)
  * Activa RC Rechargeable Neurostimulator - (Model 37612)
  * Activa SC Single Cell Neurostimulator (Models 37602 and 37603)
  * DBS Lead - (Model 3387)
  * DBS Extension - (Models 37085/6)
  * Patient Programmer - (Model 37642)
  * Test Stimulator - (Model 3625)
  * N'Vision Clinician Programmer - (Model 8840)
  * N'Vision Software Application Card - (Model 8870)
  Activa PC Primary Cell Neurostimulator - (Model 37601): Deep Brain Stimulator system will be implanted using standard neurosurgical techniques. The device will deliver constant stimulation to the thalamus using settings programmed by study team.
  Activa RC Rechargeable Neurostimulator - (Model 37612): Deep Brain Stimulator system will be implanted using standard neurosurgical techniques.
Arm/Group | DBS Active
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.5 [9 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White/ not Hispanic | 2
  White/ hispanic | 1
  other/not hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Burke-Fahn-Marsden Dystonia Rating Scale
Description: Rating scale that measures movement and disability related to dystonia, range 0-120 motor, 0-30 disability , higher number indicates more severe dystonia
  Change from Baseline in Burke-Fahn-Marsden Dystonia Rating Scale
Time Frame: Change from baseline to 12 months postoperatively
Measure: Mean (Standard Error); unit: change in points on a scale
Arm/Group | DBS Active
Number analyzed (Participants) | 4
change in points on a scale | 14.7 (11.8)

2. Primary Outcome: Percent Change in Pediatric Quality of Life Inventory (PedsQL)
Description: Quality of life measure, scored 0-100, larger scores indicate greater hinderance (ie. lower quality of life)
Time Frame: baseline to 12 months postoperatively
Measure: Mean (Full Range); unit: percent change
Arm/Group | DBS Active
Number analyzed (Participants) | 4
percent change | 27 [0 to 54.8]

3. Primary Outcome: Change in Barry Albright Dystonia Rating Scale
Description: Severity scale for secondary dystonia, range 0-32, higher scores indicates more severe dystonia
Time Frame: Change from baseline to 12 months postoperatively
Measure: Mean (Standard Error); unit: average change of points on a scale
Arm/Group | DBS Active
Number analyzed (Participants) | 4
average change of points on a scale | 0.25 (3.2)

4. Primary Outcome: Change in Blinded Burke-Fahn-Marsden Dystonia Rating Scale
Description: Rating scale that measures movement and disability related to dystonia, range 0-120 motor, 0-30 disability , higher number indicates more severe dystonia. These ratings were carried out retroactively by a neurologist who was unfamiliar with the four study participants and who had no knowledge of their unblinded scores.
Time Frame: change from baseline to 12 months postoperatively
Measure: Mean (Standard Error); unit: change in points on a scale
Arm/Group | DBS Active
Number analyzed (Participants) | 4
change in points on a scale | 4.12 (3.96)

5. Secondary Outcome: Change in Modified Ashworth Scale - Upper Limbs
Description: Measure of spasticity, range 0-32, higher values indicate more spasticity
Time Frame: Change from baseline to 12 months postoperatively
Measure: Mean (Full Range); unit: percentage change in points on a scale
Arm/Group | DBS Active
Number analyzed (Participants) | 4
percentage change in points on a scale | 0.29 [0 to 80.3]

6. Secondary Outcome: Change in Diadochokinetic Syllable Rates
Description: Articulation, range (min 6- no upper limit), longer times indicate less articulation/more difficulty with speech
Time Frame: Change from baseline to 12 months postoperatively
Population: Syllable rates collected from 2 out of the 4 participants as reported here.
Measure: Mean (Standard Deviation); unit: change in number utterances per 15 sec
Arm/Group | DBS Active
Number analyzed (Participants) | 2
change in number utterances per 15 sec | 3.25 (4.75)

7. Secondary Outcome: Children's Memory Scale
Description: Will include the following subtests: Memory for Faces, Dot Locations, and Digit Span
Time Frame: Change from baseline to 12 months postoperatively
Population: The Children's Memory Scale was not administered.
Arm/Group | DBS Active
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Behavioral Assessment System, 3rd Edition: Self Report of Personality
Description: Mood and behavior assessment, main use as a screening tool for depression.
Time Frame: Change from baseline to 12 months postoperatively
Population: Behavioral Assessment System was able to be completed by only one of the four participants. Categorical description of "atypicality" is all that was reported for the baseline and 12 month follow-up on this participant (participant 4), and no quantitative score was recorded.
Arm/Group | DBS Active
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Modified Ashworth Scale Spasticity Ratings - Lower Limbs
Description: This scale is used to measure spasticity, which is a velocity-dependent increase in muscle stretch reflexes associated with increased muscle tone as a component of upper motor neuron syndrome. It is scored 0-4 with higher scores indicating greater severity.
Time Frame: Change from baseline to 12 months postoperatively
Measure: Mean (Full Range); unit: percentage change in points on a scale
Arm/Group | DBS Active
Number analyzed (Participants) | 4
percentage change in points on a scale | 0.26 [-29.6 to 58.7]

10. Secondary Outcome: Change in Kaufman Brief Intelligence Test - Second Addition
Description: Kaufman Brief Intelligence Test Second Edition (KBIT-2) is a brief measure of verbal and nonverbal intelligence used with individuals ages 4 through 90 years, raw scores 0 - unlimited, with higher scores indicating higher ability.
Time Frame: baseline to 12 months postoperatively
Population: The Kaufman Brief Intelligence Test was only administered to 3 of the 4 participants.
Measure: Mean (Standard Deviation); unit: change BL- 12 mo. raw score on a scale
Arm/Group | DBS Active
Number analyzed (Participants) | 3
change BL- 12 mo. raw score on a scale | 6.67 (4.16)

11. Secondary Outcome: Change in Burke-Fahn-Marsden Dystonia Disability Subscale
Description: This scale is a measurement of quality of life related to dystonia, with lower scores indicating greater quality of life and high scores indicating more hinderance. It is scored 0-100.
Time Frame: baseline to 12 months postoperatively
Measure: Mean (Full Range); unit: percentage change in score on a scale
Arm/Group | DBS Active
Number analyzed (Participants) | 4
percentage change in score on a scale | 15.7 [-9.1 to 53.8]

12. Secondary Outcome: Change in Modified Unified Parkinson's Disease Rating Scale - Second Edition
Description: This scale is a measurement of quality of life related to dystonia, with lower scores indicating greater quality of life and high scores indicating more hinderance. It is scored 0-199
Time Frame: baseline to 12 months posoperatively
Population: Outcome data for this scale is only available for two of the four participants because the scale was not administered during the 12 month follow up visit for these two patients.
Measure: Mean (Full Range); unit: percentage change in points on a scale
Arm/Group | DBS Active
Number analyzed (Participants) | 2
percentage change in points on a scale | 19.25 [15 to 23.5]

ADVERSE EVENTS:
Time Frame: Patients were monitored for two years following surgery.
Arm/Group | DBS Active
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBS Active (N=4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
teeth hurt (General disorders) | 1 (1)
worsening hand movements (General disorders) | 1
drooling in sleep (General disorders) | 1 (2)
full body jerks (General disorders) | 1 (1)
fever or flu (General disorders) | 1 (1)
attitude (General disorders) | 1 (1)
viral illness (General disorders) | 1 (1)
Weight Gain (General disorders) | 1 (1)
stool incontinence (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03078816/Prot_SAP_000.pdf